CLINICAL TRIAL: NCT02062580
Title: Influence of BCG Immunization on Immune Responses and Disease Progression in South African HIV Exposed and Infected Infants
Brief Title: Early Versus Delayed BCG Vaccination of HIV-exposed Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: Seattle Children's Hospital (Other); University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Dr Heather Jaspan, Senior Lecturer, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MV-00-9-900-01871
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: HIV Exposure; HIV Infection
Keywords: Vaccine immunogenicity; Immune activation
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed BCG (Active Comparator): BCG delayed to 8 weeks of age
  Interventions: Biological: BCG
- Early BCG (Other): BCG at birth; standard of care
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: BCG

SUMMARY:
In sub-Saharan Africa (SSA), more than 300,000 babies with HIV die each year. HIV-infected children develop AIDS and die faster in SSA than those in developed countries. Bacille Calmette-Guerin (BCG) vaccine is given to infants at birth in SSA to protect them from severe forms of TB. BCG is known to cause immune cells to be active and replicate faster. The immune system of neonates also responds differently to BCG that to other vaccines and infections. We hypothesize that the routine immunization of neonates with BCG contributes to generalized immune activation in HIV-exposed infants resulting in skewed immune responses to vaccines and infections and increased rates of disease progression in those infants that become HIV-infected. However, delaying BCG until HIV testing is completed would result in operational difficulties, and may not induce the appropriate immune response. Delayed BCG would also render many HIV-exposed uninfected infants at high risk for disseminated TB. We plan to assess immune cells in infants to determine the impact of the timing of BCG vaccination on immune responses to tuberculosis (TB) and other vaccines. We will also compare the immune activation and disease progression of those infants that become HIV-infected in the BCG or control arms. Our results will provide key insights into the effect of BCG vaccination on immune responses to HIV as well as inform the optimal timing of BCG vaccination for HIV-exposed infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy neonate
* Maternal HIV
* > 36 weeks gestation
* Birth weight > 2.4kg
* Remaining in area 4 months

Exclusion Criteria:

* Complications during pregnancy and delivery
* Household TB contacts

Max Age: 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 149 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather B Jaspan, MD, PHD, Principal Investigator — University of Cape Town

REFERENCES:
- [Derived] Gasper MA, Hesseling AC, Mohar I, Myer L, Azenkot T, Passmore JS, Hanekom W, Cotton MF, Crispe IN, Sodora DL, Jaspan HB. BCG vaccination induces HIV target cell activation in HIV-exposed infants in a randomized trial. JCI Insight. 2017 Apr 6;2(7):e91963. doi: 10.1172/jci.insight.91963. PMID 28405623
- [Derived] Blakney AK, Tchakoute CT, Hesseling AC, Kidzeru EB, Jones CE, Passmore JA, Sodora DL, Gray CM, Jaspan HB. Delayed BCG vaccination results in minimal alterations in T cell immunogenicity of acellular pertussis and tetanus immunizations in HIV-exposed infants. Vaccine. 2015 Sep 11;33(38):4782-9. doi: 10.1016/j.vaccine.2015.07.096. Epub 2015 Aug 7. PMID 26259542
- [Derived] Tchakoute CT, Hesseling AC, Kidzeru EB, Gamieldien H, Passmore JA, Jones CE, Gray CM, Sodora DL, Jaspan HB. Delaying BCG vaccination until 8 weeks of age results in robust BCG-specific T-cell responses in HIV-exposed infants. J Infect Dis. 2015 Feb 1;211(3):338-46. doi: 10.1093/infdis/jiu434. Epub 2014 Aug 8. PMID 25108027

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed BCG: BCG delayed to 8 weeks of age
  BCG
- Early BCG: BCG at birth; standard of care
  BCG
Period: Overall Study
Arm/Group | Delayed BCG | Early BCG
Started | 71 | 78
Completed | 59 | 65
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Delayed BCG | Early BCG | Total
Number analyzed (Participants) | 71 | 78 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 71 | 78 | 149
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Median gestational age, in weeks
  weeks | 39 [38 to 40] | 40 [39 to 40] | 39.5 [38 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 46 | 87
  Male | 30 | 32 | 62
Region of Enrollment [Number; unit: count of participants]
  South Africa | 70 | 76 | 146
Birth weight [Median (Inter-Quartile Range); unit: kg] | 3.15 [2.85 to 3.3] | 3.12 [2.8 to 3.4] | 3.13 [2.9 to 3.4]
Maternal CD4 T cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 358 [254 to 548] | 366 [271 to 477] | 362 [263 to 513]
Breastfed [Number; unit: participants]
  yes | 8 | 12 | 20
  no | 62 | 64 | 126

OUTCOME MEASURES:

1. Primary Outcome: T Cell Activation
Description: Percentage of all CD4+ T cells expressing HLADR (NOT BCG-specific activation as in Tchakoute et al and as in secondary outcome). The n is smaller than the enrollment number as some participants were lost to follow-up, some were excluded due to HIV infection etc, and some samples did not have sufficient cells to analyse.
Time Frame: at 6 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of CD4+ T cells
Arm/Group | Delayed BCG | Early BCG
Number analyzed (Participants) | 63 | 68
percentage of CD4+ T cells | 1.8 [1 to 2.8] | 1.3 [0.8 to 2.4]

2. Secondary Outcome: Vaccine Immunogenicity
Description: Percent of CD4+ T cells expressing Ki67 after stimulation in vitro with BCG.
Time Frame: 6 weeks after BCG vaccination
Population: Analysis population n is smaller than enrollment numbers as we calculated that that only 28 were needing in each arm to detect a difference.
Measure: Median (Inter-Quartile Range); unit: percentage of Ki67% CD4+ T cells
Arm/Group | Delayed BCG | Early BCG
Number analyzed (Participants) | 28 | 28
percentage of Ki67% CD4+ T cells | 22.4 [4.7 to 28.5] | 20.5 [10 to 31.5]

ADVERSE EVENTS:
Arm/Group | Delayed BCG | Early BCG
Serious Adverse Events (participants affected / at risk) | 2/71 | 7/78
Other Adverse Events (participants affected / at risk) | 29/71 | 30/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed BCG (N=71) | Early BCG (N=78)
HIV infection (Immune system disorders) | 2 (2) | 4
Death (General disorders) | 0 (0) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Delayed BCG (N=71) | Early BCG (N=78)
Blocked nostrils (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 11 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 15 (15)
Fever (General disorders) | 6 (6) | 6 (6)
Rash- nonspecific (Skin and subcutaneous tissue disorders) | 9 (9) | 10 (10)
Diaper Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No